CLINICAL TRIAL: NCT05321225
Title: The Level of Blood Brain Barrier Damage Biomarker Predicting Hemorrhagic Transformation Following Acute Ischemic Stroke
Brief Title: The Level of Blood Brain Barrier Damage Biomarker in Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor of Neurosurgery, Vice-President of Xuan Wu Hospital, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: BBBD-AIS
Record Dates: First submitted 2022-03-19; First posted 2022-04-11 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Stroke
Keywords: blood brain barrier; hemorrhagic transformation; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood samples from enrolled patients on admission was drawn by emergency department nurse using containing coagulant tubes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: the level of biomarker in bood — Elisa is used to test the level of biomarker in blood.

SUMMARY:
Hemorrhagic transformation is a common complication of acute ischemic stroke patients . BBB damage is regarded as a major pathophysiological mechanism of hemorrhagic transformation. So, the investigators hypothesis the level of BBB damage biomarker is predictor of intracranial hemorrhage following ischemic stroke.

DETAILED DESCRIPTION:
Hemorrhagic transformation is a common complication of acute ischemic stroke patients . BBB injury often occurs in the early stage of ischemic stroke, leading brain tissue edema or even hemorrhagic transformation with the development of ischemic injury. The biomarker of BBB damage, such as the level of serum occludin, can reflect the extent of BBB injury. So, the investigators hypothesis the level of BBB damage biomarker is predictor of intracranial hemorrhage following ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled patients aged 18-80years.
2. Acute ischemic stroke
3. Informed consent obtained.

Exclusion Criteria:

1. Tumor stroke or hemorrhagic stroke or hemorrhagic cerebral infarction on admission.
2. Stroke or serious head trauma within the previous 3 months
3. inflammatory or infectious diseases, cancer, coagulation disturbance disease and severe renal and liver failure
4. blood sample occurred hemolysis or cloudy.
5. Incomplete clinical data
6. Platelet count of less than 100,000 per cubic millimeter
7. Received oral anticoagulation therapy preceding the onset of stroke and INR greater than 1.7 or prothrombin times greater than 15 seconds
8. Pregnant or breast-feeding women
9. Patients being enrolled or having been enrolled in other clinical trial -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients received standard therapy within 24-hour since stroke onset
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of serum biomarkers within 72h in ischemic stroke patients | Day 0, Day 1, Day 2, Day 3.
  The level of biomarkers are detected using Elisa(Enzyme Linked Immunosorbent Assay)，biomarkers including Occludin(ng/mL), Claudin-5(ng/mL), MMP-2/9(ng/mL)，c-Fn(ug/mL), ZO-1(pg/mL), vWF(ng/mL), IL-2RA(ng/mL), CCL16(ng/mL), CNTN(ng/mL), SELE(ng/mL) and PGLYRP1(ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Ke Jian Liu, PhD, Principal Investigator — Xuan Wu Hospital,Capital Medical University
Locations (1):
- Xuanwu hospital;Capital Medical University, Beijin, XI Cheng District, China

IPD SHARING:
Plan to Share IPD: Yes